CLINICAL TRIAL: NCT00036608
Title: A Phase III Study of Entecavir vs Lamivudine in Chronic Hepatitis B Subjects With Incomplete Response to Lamivudine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Purpose: Treatment
Other Study IDs: AI463-026
Record Dates: First submitted 2002-05-10; First posted 2002-05-13 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2010-01

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir

INTERVENTIONS:
Drug: Entecavir

SUMMARY:
The purpose of this clinical research study is to assess the safety and effectiveness of switching to entecavir compared to continued lamivudine in patients with chronic hepatitis B.

ELIGIBILITY:
* Male and female subjects =/> 16 years of age (or minimum age required in a given country) with history of HBeAg-positive chronic hepatitis B infection;
* Incomplete response to current lamivudine therapy;
* HBeAg-positive;
* Absence of coinfection with human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis D virus (HDV);
* Absence of other forms of liver disease e.g., alcoholic, autoimmune, biliary disease.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-01; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (34):
- United States (34):
  - Local Investigator, Birmingham, Alabama
  - Local Investigator, Tucson, Arizona
  - Local Investigator, La Jolla, California
  - Local Investigator, Los Angeles, California
  - Local Investigator, Orange, California
  - Local Investigator, San Diego, California
  - Local Investigator, San Francisco, California
  - Local Investigator, Farmington, Connecticut
  - Local Investigator, Miami, Florida
  - Local Investigator, Miami Beach, Florida
  - Local Investigator, Atlanta, Georgia
  - Local Investigator, Honolulu, Hawaii
  - Local Investigator, Chicago, Illinois
  - Local Investigator, Iowa City, Iowa
  - Local Investigator, New Orleans, Louisiana
  - Local Investigator, Dundalk, Maryland
  - Local Investigator, Boston, Massachusetts
  - Local Investigator, Worcester, Massachusetts
  - Local Investigator, Ann Arbor, Michigan
  - Local Investigator, Royal Oak, Michigan
  - Local Investigator, Saint Paul, Minnesota
  - Local Investigator, Manhasset, New York
  - Local Investigator, New York, New York
  - Local Investigator, Rochester, New York
  - Local Investigator, Charlotte, North Carolina
  - Local Investigator, Durham, North Carolina
  - Local Investigator, Cleveland, Ohio
  - Local Investigator, Philadelphia, Pennsylvania
  - Local Investigator, Pittsburgh, Pennsylvania
  - Local Investigator, Providence, Rhode Island
  - Local Investigator, Nashville, Tennessee
  - Local investigator, Dallas, Texas
  - Local Investigator, Fairfax, Virginia
  - Local Investigator, Richmond, Virginia